## STATISTICAL ANALYSIS PLAN

## LIPID-LOWERING REGIMES IMPROVE OXIDATIVE STRESS, TRYPTOPHAN DEGRADATION IN HYPERCHOLESTEROLEMIA CKD PATIENTS

Date of review: 05th May, 2018

All results will be expressed as mean values (mean SD) or median values (median and range).

The statistical differences between the mean laboratory test results patients and control group will be analyzed by ANOVA one-way statistical analysis or by Student's t-test (with Kolmogorov-Smirnov for normality).

The statistical differences in the effect of each therapy on laboratory mean values will be evaluated by one way repeated measure ANOVA with Bonferroni correction or Dunnet T3 correction, if appropriate.

To compare the differences in the median values of laboratory tests between 3 groups, ANOVA one-way will be applied. If there are statistical differences between 3 groups, we will use deeply ANOVA one-way test to analyze which group is different from another group (with Bonferroni if Levene test  $\geq 0.05$  or Dunnet T3 if Levene test < 0.05).

Correlation analysis between variables will be performed by Pearson's correlation or Spearman's correlation as appropriate.

Statistical analysis will be performed by using SPSS for Windows, version 20.0 (IBM Corporation; Armonk, NY, USA).